CLINICAL TRIAL: NCT01159418
Title: A Phase IB Study of the Histone Deacetylase Inhibitor Panobinostat (LBH589) Given Orally in Combination With Carboplatin and Paclitaxel in Patients With Advanced Solid Tumors
Brief Title: LBH589 Oral in Combination With Carboplatin and Paclitaxel in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southern Europe New Drug Organization (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKSD00702
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Advanced Solid Tumors
Keywords: solid tumors; Panobinostat; histone deacetylase inhibitors
MeSH Terms: interventions — Panobinostat; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panobinostat (LBH589), Carboplatin and Paclitaxel (Experimental)
  Interventions: Drug: Panobinostat (LBH589), Carboplatin and Paclitaxel

INTERVENTIONS:
Drug: Panobinostat (LBH589), Carboplatin and Paclitaxel — 1. Panobinostat (LBH589) p.o. on days 1,4,8 and 11 of each cycle (20mg-45mg).Carboplatin i.v.on day 1 at a total dose corresponding to a AUC of 5 µg/ml.h. Paclitaxel as 3 hour infusion on day 1 (135 mg/m2).
  2. Panobinostat (LBH589) p.o. on days 1, 4, 15 and 18 of each cycle (20mg-30mg).Carboplatin i.v. on day 8 at a total dose corresponding to a AUC of 5 µg/ml.h.Paclitaxel as a 3 hour infusion on day 8 (135mg/m2-175mg/m2).
  3. Once the MTD is achieved:Panobinostat (LBH589) p.o. on days 1 and 4 of each cycle(20mg-30 mg). Carboplatin i.v. on day 8 at a total dose corresponding to a AUC of 5 µg/ml.h.Paclitaxel as a 3 hour infusion on day 8 (135mg/m2-175 mg/m2).
  The treatment will be repeated every three weeks until disease progression.

SUMMARY:
The purpose of this study is to determine the Maximum Tolerated Dose (MTD) of Panobinostat (LBH589) when administered in combination with Carboplatin and Paclitaxel in patients with advanced solid malignancies and to identify the Recommended Dose (RD) for a subsequent Phase II study.

DETAILED DESCRIPTION:
The combination of Carboplatin (C) and Paclitaxel (PTX) is considered standard treatment in patients with epithelial ovarian cancer and endometrial cancer, in USA and in those in whom anthracyclines are not recommended. In cervical cancer, where very often the renal function is impaired, C represents a convenient substitute of cisplatin in the combination with PTX; in NSCLC the C and PTX regimen is first choice therapy for outpatient treatment first or second line.

LBH is a histone deacetylase (HDAC) inhibitor available also for oral administration.

In combination with platinum agents LBH589 could improve efficacy on DNA by multiple non-exclusive mechanisms (by increasing drug access to chromosomal DNA, interfering with DNA repair, modulating the levels of pro antiapoptotic genes or proliferation/survival genes).

The inclusion of Paclitaxel in the combination of LBH589 and Carboplatin is supported by the results already available with the combination of the HDAC inhibitor Vorinostat (suberoylanilide hydroxamic acid) given orally with carboplatin (AUC 6 mg/ml.h) and paclitaxel (200 mg/m2) in a Phase I study in patients with solid tumors. The regimen proved to be feasible, well tolerated and was associated with promising antitumor activity in patients with NSCLC.

The mechanism of action, and the preliminary preclinical data, suggest that the combination of LBH589, Carboplatin and Paclitaxel could be feasible and worthy of clinical investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Histological/cytological diagnosis of solid tumors in which treatment with Carboplatin and Paclitaxel is indicated, e.g. NSCLC, GY tumors, prostate cancer, unknown primary
2. Progressive disease (also in terms of tumor markers only, like CA 125 for ovary and PSA for prostate).
3. Age 18-75 years
4. Prior chemotherapy of ≤ 1 line for advanced disease
5. ECOG Performance Status < 2
6. Life expectancy of at least 3 months
7. The patient must be able to read, understand and provide written evidence of informed consent
8. Female patients may not be pregnant or lactating and must be willing to practice contraception. The effects of LBH589 on the developing human fetus are unknown. For this reason, women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation.
9. Male patients that are not surgically sterile must be practicing a medically acceptable contraceptive regimen while on study treatment
10. Adequate organ function as defined by the following:

    * ANC > 1500/µL
    * Platelets ≥ 100,000/µL
    * Haemoglobin ≥ 10 g/dl
    * Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 60 ml/min
    * Magnesium, potassium and phosphorus ≥ the lower limit of normal or correctable with supplements
    * Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) ≤ 2.5 x ULN or ≤ 5.0 x ULN if hepatic involvement is present
    * Serum bilirubin ≤ 1.5 x ULN
    * Alkaline phosphatase (ALP) ≤ 2.5 x ULN or ALP > 2.5 x UNL with liver fraction ≤ 2.5 x ULN

Exclusion Criteria:

1. Other chemotherapy treatment < 4 weeks prior to enrolment
2. Hypersensitivity or allergic reactions to platinum compounds or Carboplatin®; hypersensitivity or allergic reactions to Paclitaxel
3. Radiotherapy involving > 30% of the active bone marrow
4. Radiotherapy < 4 weeks prior to enrolment
5. Pre-existing peripheral neuropathy ≥ grade 2
6. Pre-existing CTCAE hearing loss or tinnitus ≥ grade 2
7. Symptomatic pleural effusion
8. Clinically significant third space fluid accumulation (e.g. ascites,..)
9. Symptomatic brain metastasis or meningeal tumors
10. Patients who have not recovered (> grade 1) from the following toxicities of previous regimens before enrolment: fatigue, mucositis, nausea/vomiting, diarrhea
11. Concurrent enrolment, or previous enrolment within 30 days prior to registration in another investigational device or drug trial(s) or is receiving other investigational agent(s)
12. Human immunodeficiency virus (HIV) infection
13. History of bone marrow or major organ transplant
14. Prior high dose treatment with PBSC support
15. Impaired cardiac function, including any one of the followings:

    * Complete Left Bundle Branch Block or obligate use of a cardiac pacemaker or congenital long QT syndrome or history or presence of atrial or ventricular tachyarrhythmias or clinically significant resting bradycardia (< 50 beats per minute) or QTcF > 480 msec on screening ECG or Right Bundle Branch block + left anterior hemiblock (bifascicular block)
    * Angina pectoris or acute MI ≤ 3 months prior to starting study drug
    * Other clinically significant heart disease (e.g. congestive heart failure, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
16. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral LBH589 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, malabsorption syndrome, or small bowel resection)
17. Acute or chronic liver or renal disease
18. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes, active or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease) that could cause unacceptable safety risks or compromise compliance with the protocol
19. Concomitant use of CYP3A4/5 inhibitors or inducers where the treatment can not be discontinued or switched to a different medication prior to starting study drug (medications listed in Appendix 3). The medications listed in Appendix 3 have a relative risk of prolonging the QT interval or inducing Torsades de Pointes, but do not represent an exclusion criteria
20. Treatment with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GMCSF) ≤ 2 weeks prior to starting study drug.
21. Treatment with therapeutic doses of sodium warfarin (Coumarin ). Low doses of Coumarin (e.g., ≤ 2 mg/day) for line patency is allowable
22. Patients who have received biologic therapy (excluding antiangiogenics) or immunotherapy ≤ 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy
23. Patients who have undergone major surgery ≤ 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
24. Unable or unwilling to comply with all study procedures
25. Current history of alcohol or drug abuse

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-12 (Estimated); Study Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) Recommended Dose (RD) | 3 weeks after the first drug administration (1 Cycle)
  Number of Dose-Limiting Tocixities (DLTs)

SECONDARY OUTCOMES:
Hints of antitumor activity | from first drug administration until tumor progression (every 6 weeks)
  objective tumor responses based on RECIST criteria
Biomarkers of HDAC | Cycle 1 on day 1, 4, 8, 15 and Cycle 2 on day 1, 8.
  acetylation of histones, H3, H4 and tubulin in PBMC
Safety and tolerability | 4 weeks after last drug administration
  AE types and frequency monitored by laboratory and instrumental assessments, and physical examination

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - Huniversitätsspitals Basel, Basel
  - Istituto Oncologico della Svizzera Italiana, Bellinzona
  - Mèdecin Adjoint, ME - CePO, CHUV, Lausanne